CLINICAL TRIAL: NCT05405101
Title: A Prospective Randomised Trial Comparing Thermal Ablation With Laparoscopic Adrenalectomy as an alternatiVE Treatment for Unilateral Asymmetric Primary Aldosteronism
Brief Title: Randomised Trial Comparing Thermal Ablation With Adrenalectomy in the Treatment of Unilateral Asymmetric PA
Acronym: WAVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 304174
Record Dates: First submitted 2022-03-15; First posted 2022-06-06 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Primary Aldosteronism
Keywords: Thermal; Ablation; Laparoscopic; Adrenalectomy
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Intervention Model Description: PROBE: Prospective Randomised open blinded end point study. Patients are randomized using a minimization program. 2:3 Surgery: Ablation
Who Masked: Outcomes Assessor
Masking Description: PROBE (Prospective, Randomised, Open-label with Blind Endpoint) multi-centre comparison of thermal ablation with laparoscopic adrenalectomy in the treatment of unilateral asymmetric primary aldosteronism.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thermal ablation of adrenal aldosterone producing adenoma (s) (Experimental): For patients randomized to ablation, thermal ablation (either microwave or radiofrequency ablation) will be deployed to treat the adrenal aldosterone producing adenoma(s)
  Interventions: Procedure: Thermal ablation of aldosterone producing adenoma.
- Unilateral adrenalectomy for aldosterone producing adenoma (s) (Other): For patients randomized to surgery, unilateral adrenalectomy will be performed to remove aldosterone producing adenoma(s)
  Interventions: Procedure: Unilateral adrenalectomy

INTERVENTIONS:
Procedure: Thermal ablation of aldosterone producing adenoma. — On the left side, Radiofrequency ablation of aldosterone producing adenoma(s) will be undertaken via the stomach (endoscopically), under transgastric ultrasound guidance.
  On the right side, either Radiofrequency or Microwave Ablation of aldosterone producing adenoma(s) will be performed via a percutaneous approach, under CT guidance.
  Arms: Thermal ablation of adrenal aldosterone producing adenoma (s)
Procedure: Unilateral adrenalectomy — Unilateral total adrenalectomy for aldosterone producing adenoma. This will be laparoscopic in the vast majority of patients, with open conversion if surgically indicated (unlikely in >1-2 patients)
  Other Names: Laparoscopic adrenalectomy
  Arms: Unilateral adrenalectomy for aldosterone producing adenoma (s)

SUMMARY:
The primary objective of WAVE is to test the hypothesis that thermal ablation (microwave or RFA) is non-inferior to surgery in the biochemical (and if so, in the clinical) cure of unilateral PA, according to the international consensus PASO criteria.

Secondary objectives are to determine whether either intervention is superior to the other in relation to the following outcomes. Where no superiority of either intervention is established, non-inferiority of thermal ablation against adrenalectomy will be sought.

* Frequency and severity of adverse events
* Length of inpatient stay
* Patient satisfaction
* Quality of life
* Return to activities of daily living

An additional secondary objective in the thermal ablation group alone will be anatomical efficacy of ablation.

DETAILED DESCRIPTION:
Primary aldosteronism (PA) results from renin-independent aldosterone hypersecretion and causes hypertension, often with associated hypokalaemia and metabolic alkalosis. These are due to enhanced mineralocorticoid receptor-mediated renal sodium retention and potassium excretion. PA is the commonest cause of secondary hypertension and is responsible for 5-10% of all hypertension, rising to in excess of 20% of resistant cases. Very low diagnosis rates result from a generation of doctors schooled on order-of-magnitude lower estimates, but recent findings suggest that even the 5-10% prevalence may be a considerable under-estimate. In addition to its frequency, PA is a high-risk subset of hypertension and is associated with a two-fold increased risk of cardiovascular events and atrial fibrillation compared to comparable patients with essential hypertension, as well as a reduced quality of life.

Aldosterone excess in PA can originate from one or both adrenal glands. Patients with PA are considered to divide ~50:50 into those with a curable unilateral aldosterone-producing adenoma (APA), and those with bilateral idiopathic adrenal hyperplasia (IAH). For patients with unilateral PA, surgical removal of the affected gland (adrenalectomy) is highly likely to cure the biochemical abnormality, reverse the excess cardiovascular and stroke risks, and is strongly supported by international guidelines.

Whilst directed medical therapies against aldosterone excess exist (e.g. mineralocorticoid receptor antagonists, MRAs), they are inferior to surgery in reducing the excess cardiovascular and stroke risk and improving quality of life. Furthermore, sufficient MRA dosing to de-suppress renin and reverse this excess risk is only achieved in one-third of medically-treated patients. The case for definitive intervention in unilateral PA is therefore compelling, and recommended whenever possible. At present, this is achieved by laparoscopic adrenalectomy (LA), which involves a general anaesthetic, inpatient admission and removal of the entire adrenal gland to treat a condition caused by a small (usually <2cm diameter, often <1cm) benign APA.

An alternative intervention to LA, and the focus of this trial, is selective thermal ablation (by radiofrequency or microwave) of the identified APA(s). Thermal ablation is a technique in which targeted and directed tissue death can be achieved with precision under image guidance, sparing the normal adrenal gland. It is widely established in the treatment of benign and malignant hepatic and renal neoplasms as an alternative to conventional surgery. For these indications, thermal ablation techniques have transformed practice, not only providing high-risk surgical patients with a previously unobtainable curative treatment option but also becoming an accepted mainstay of treatment for small lesions (of the size encountered in PA) in all patients regardless of surgical risk.

We propose a multi-centre prospective randomised trial comparing adrenalectomy (LA) and thermal ablation for the treatment of unilateral APAs. This study is powered to demonstrate non-inferiority of biochemical and clinical response to thermal ablation, compared to the current standard of care, adrenalectomy. The rationale for a non-inferiority trial is that subsequent preference for thermal ablation over surgery will be driven by thermal ablation's greater patient-acceptability and availability, rather than an implausible superior efficacy of sub-total than total adrenalectomy in curing PA. Once safety and efficacy are proven as comparable to those of adrenalectomy, thermal ablation has potential for superiority over medical treatment in several patient groups ineligible for WAVE, e.g., some with bilateral disease, or in whom lateralisation could not be performed.

ELIGIBILITY:
Inclusion criteria (all of):

* Age > 18 years
* Primary aldosteronism diagnosed according to international guidelines
* Unilateral disease by AVS or PET-CT criteria
* Ipsilateral radiological abnormality with benign imaging characteristics and technically amenable to both thermal ablation and surgery
* Able and willing to give informed consent
* Randomisation approved by MDT

Exclusion criteria (any of):

* Absolute contraindication to α- or β-adrenoceptor antagonist therapy or CT contrast
* Contraindication or unwillingness for either surgery or thermal ablation
* Inability to withdraw β-adrenoceptor antagonist therapy for 2 weeks
* Unwilling to undergo either LA or thermal ablation
* Unwilling to comply with study visit schedule
* Pregnancy or unwillingness to undertake secure contraception for the study duration (female participants only)
* Life-limiting comorbidity (at the discretion of the PI)
* Clinical and/or biochemical evidence of autonomous cortisol secretion sufficient, in the opinion of the patient's physician, to mandate a unilateral adrenalectomy independent of autonomous aldosterone secretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Complete biochemical cure of PA | 6 months post intervention
  Complete biochemical cure of PA, defined (whilst off medications that might alter serum potassium or the RAS) by both:
  1. Normalisation of serum potassium, and
  2. Normalisation of ARR, or
  3. Elevated ARR and
  i. Baseline PAC <190pmol/L, or ii. Normal confirmatory test (as defined in the inclusion criteria)
Complete clinical cure of PA | 6 months post intervention
  Complete clinical cure of PA, defined as normotension without antihypertensive medication
  These criteria have been defined in the international consensus PASO statement8, which has become the established yardstick by which PA cure is judged. In this, normotension is defined, in accordance with the European Society of Hypertension guidelines22, as <140/80 in the office, <135/85 at home or daytime ambulatory monitoring and <130/80 for 24h ambulatory blood pressure monitoring (24hABPM).

SECONDARY OUTCOMES:
Adverse events | Reported throughout the study period. Approximately 2 years
  * Will be directly sought at each study visit through history and physical examination where appropriate
  * Subjects will be encouraged to report between study visits and will have a mechanism to do so
  * Will be classified by system, seriousness, causal relationship and expectedness according to the Common Terminology Criteria for Adverse Events v5.0 (CTCAE)
Anaemia (FBC, requirement for blood transfusion) | 6, 12, 24 and 36 months post intervention
  Blood test
Renal dysfunction and electrolyte abnormalities (U&Es) | 6, 12, 24 and 36 months post intervention
  Blood test
Liver dysfunction (LFTs) | 6, 12, 24 and 36 months post intervention
  Blood test
Pancreatitis (lipase/amylase) | 6, 12, 24 and 36 months post intervention
  Blood test
Hypertensive urgency (physiological parameters, plasma metanephrines) | 6, 12, 24 and 36 months post intervention
  Blood test
Length of inpatient stay (hospital episode data) | 6 weeks post intervention
  As reported by patient
Patient satisfaction (Freiburg index of patient satisfaction) | 6 weeks post intervention
  Completed by patient, using the FIPs score values to rate the treatment they have received.
Quality of life questionnaire | 6 months post intervention
  Completed by patient, using the - EQ-5D 5L and SF-36 questionnaire models to score self rated health and quality of life values. These 2 models are presented as one questionnaire to the patient.
Return to usual activities of daily living (self-reported) | 6 weeks post intervention
  As reported by patient
Anatomical efficacy of ablation | 6, 12, 24 and 36 months post intervention
  (ablation group only; post-ablation Metomidate/CETO PET-CT appearances)

OTHER OUTCOMES:
Hierarchical analysis testing | 6 months post intervention
  Hierarchical analysis testing will be applied to sequential testing of the following hypotheses. Each positive outcome permits the next limb to be tested as a co-primary hypothesis. A negative outcome converts subsequent limbs to secondary hypotheses.
  [i] Complete biochemical cure for left ablation vs left surgery (positive if non-inferiority (NI) margin <45%) [ii] Complete biochemical cure for all ablation vs all surgery (positive if NI margin <45%) [iii] Complete clinical cure for all ablation vs all surgery (positive if NI margin <33%) The first limb of the hierarchy will be tested if sufficient patients have been recruited on the left, anticipated to be 3 times as many as on the right.

CONTACTS AND LOCATIONS:
Overall Officials: Morris Brown, Principal Investigator — Queen Mary University of London
Locations (6):
- United Kingdom (6):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge, SMLG
  - St Bartholomew's Hospital, London
  - University College London Hospital NHS Foundation Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: Undecided
Once discussed with patient representative from patient and public Involvement, document will be uploaded on to system following first Trial Steering Committee involving PPI member